CLINICAL TRIAL: NCT04185363
Title: An Open-label Extension Study to Evaluate the Long-term Safety and Efficacy of Maralixibat in the Treatment of Subjects With Progressive Familial Intrahepatic Cholestasis (PFIC)
Brief Title: An Extension Study of Maralixibat in Patients With Progressive Familial Intrahepatic Cholestasis (PFIC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRX-503
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Progressive Familial Intrahepatic Cholestasis (PFIC)
Keywords: Cholestasis; Maralixibat; Mutation; PFIC; PFIC2; Bile Duct Diseases; Liver Diseases; Biliary Tract Diseases; Digestive System Diseases; Pediatric
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1; Cholestasis; Bile Duct Diseases; Liver Diseases; Biliary Tract Diseases; Digestive System Diseases | interventions — maralixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Maralixibat (Experimental): All subjects will receive Maralixibat oral solution
  Interventions: Drug: Maralixibat

INTERVENTIONS:
Drug: Maralixibat — All subjects will receive Maralixibat oral solution (up to 600 microgram per kilogram [mcg/kg]) twice daily

SUMMARY:
The primary objective of this open label extension study is to evaluate the long-term safety and tolerability of maralixibat.

DETAILED DESCRIPTION:
The study will be conducted at multiple sites in North America, Europe, Asia, and South America.

ELIGIBILITY:
Key Inclusion Criteria:

1. Provide informed consent and assent (as applicable) per Institutional Review Board/Ethics Committee (IRB/EC)
2. Completion of study MRX-502

Exclusion Criteria:

1. Any female who is pregnant or lactating or who is planning to become pregnant
2. Administration of prohibited medication between the MRX-502 EOT visit and the MRX 503 Baseline Visit (Day 0)
3. History of non-compliance in study MRX-502, non-adherence to medical regimens, unreliability, mental instability or incompetence that could compromise the validity of informed consent or lead to non-adherence with the study protocol based on Investigator judgment
4. Experienced an adverse event (AE) or serious adverse event (SAE) related to maralixibat during the MRX-502 study that led to permanent discontinuation of the subject from maralixibat
5. Any other conditions or laboratory abnormalities that, in the opinion of the Investigator or Sponsor Medical Monitor, may compromise the safety of the subject, or interfere with the subject participating in or completing the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) during the study | From baseline through time of interim analysis, up to 120 weeks

SECONDARY OUTCOMES:
Change from maralixibat baseline over the course of the study in the weekly average morning ItchRO(Obs)™ (Itch Reported Outcome) severity score | From baseline through study completion, up to approximately 4 years
Maintenance of treatment effect based on the average morning ItchRO(Obs)™ severity scores over the time | From baseline through study completion, up to approximately 4 years
Mean change from baseline over time in serum bile acid (sBA) levels | From baseline through study completion, up to approximately 4 years
Change from maralixibat baseline over the course of the study in the weekly average morning ItchRO(Obs)™ (Itch Reported Outcome) frequency score | From baseline through study completion, up to approximately 4 years
Mean change from baseline over time in height and weight z-scores | From baseline through study completion, up to approximately 4 years

CONTACTS AND LOCATIONS:
Locations (28):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Advent Health, Orlando, Florida
  - Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas, Health Science Center San Antonio, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Medizinische Universität Wien, Universitätsklinik für Kinder- und Jugendheilkunde, Vienna, Austria
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Sociedade Beneficente de Senhoras Hospital Sírio-Libanês, São Paulo, Brazil
- University of Alberta - Women and Children's Health Research Institute, Edmonton, Alberta, Canada
- Fundacion Cardioinfantil, Bogotá, Colombia
- France (2):
  - Groupement Hospitalier Est Hopital, Femme Mère Enfant de Lyon, Lyon
  - CHU de Toulouse - Hôpital des Enfants, Toulouse
- Medizinische Hochschule, Hanover, Germany
- Italy (2):
  - Azienda Ospedaliera Papa Giovanni XXIII - Unita di Pediatria, Bergamo
  - Ospedale Pediatrico bambino Gesu', Roma
- Hotel Dieu de France, Alfred Naccache, Beirut, Lebanon
- Consultario de Joshue David Covarrubias Esquer, Zapopan, Mexico
- Instytut Pomnik Centrum, Zdrowia Dziecka, Warsaw, Poland
- KK Women's and Children's Hospital, Singapore, Singapore
- Koc University Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Genetics Home Reference - PFIC — https://ghr.nlm.nih.gov/condition/progressive-familial-intrahepatic-cholestasis
- See also: US FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks
- See also: Mirum Pharmaceuticals homepage — https://mirumpharma.com/